CLINICAL TRIAL: NCT00586989
Title: Endoscopic Tri-Modal Imaging for the Detection of High-Grade Dysplasia and Early Adenocarcinoma in Patients With Barrett's Esophagus: A Randomized Crossover Multi-center Study
Brief Title: Endoscopic Tri-Modal Imaging in Patients With Barrett's Esophagus
Acronym: ETMI
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Louis-Michel Wong Kee Song, Principal Investigator, Mayo Clinic
Other Study IDs: 07-003997; 07-003997
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2010-09

CONDITIONS: Barretts Esophagus; High Grade Dysplasia; Early Esophageal Adenocarcinoma
Keywords: Barrett's Esophagus; Esophageal Cancer; High Grade Dysplasia
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus; Esophageal Neoplasms | interventions — Gastroscopy; Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — esophageal biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patient with Barrett's Esophagus with a history of High grade dysplasia or early esophageal adenocarcinoma
  Interventions: Procedure: Upper endoscopy with biopsy

INTERVENTIONS:
Procedure: Upper endoscopy with biopsy — Endoscopy with biopsy 6 weeks after the initial endoscopy
  Other Names: ETMI system (Olympus, Tokyo, Japan)

SUMMARY:
This study is being done to determine if a new endoscope will help doctors identify pre-cancer or early cancer lesions in patients who have Barrett's esophagus. This new endoscope allows the doctor to look at the lining of the esophagus in 3 different ways by modifying light.

DETAILED DESCRIPTION:
Patients with Barrett's esophagus are advised to undergo periodic endoscopic surveillance with random biopsies in an attempt to identify high-grade dysplasia (HGD) or early adenocarcinoma (ACA) at a time when intervention can be curative. This approach, however, can be time-consuming and is hindered by low sampling yield and random sampling error. Endoscopic Tri-Modal Imaging (ETMI) is a novel diagnostic modality that encompasses three advanced imaging features in one system: high-resolution endoscopy (HRE), autofluorescence imaging (AFI) and narrow-band imaging (NBI). HRE and AFI provide a bird's-eye view of 'red flag' areas which are then assessed by NBI for focused and more specific tissue characterization. The aim of this prospective, multi-center study is to compare the diagnostic performance of ETMI with that of standard white-light endoscopy (WLE) for identifying high-grade dysplasia (HGD) and early adenocarcinoma (ACA) in BE. A total of 84 BE patients will be recruited for the study and they will undergo both ETMI and WLE examinations in a randomized, crossover fashion. Standard surveillance biopsies and ETMI-targeted biopsies will be performed. The primary outcome will compare the number of patients and lesions with HGD or early ACA detected with WLE and ETMI. It is anticipated that ETMI will enhance the detection of high-grade Barrett's lesions relative to WLE.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Prior diagnosis of BE, defined as the presence of columnar-lined epithelium in the distal tubular esophagus with specialised intestinal metaplasia on histological investigation
3. Prior diagnosis of HGD or early ACA that was endoscopically inconspicuous according to the referring source
4. A minimum Barrett's length of C>2M>2 or C<2M>4 according to the Prague C&M classification for the endoscopic appearance of BE
5. Ability to provide written informed consent

Exclusion Criteria:

1. Description of a visibly suspicious lesion within the Barrett's segment according to the referring source
2. Presence of a type 0-I or type 0-III lesion, or a lesion that, according to the discretion of the endoscopist, does not allow delay in intervention for a period of 6 weeks (minimum interval between the two crossover endoscopies)
3. Prior endoscopic therapy for Barrett's lesions, such as photodynamic therapy or endoscopic mucosal resection (EMR)
4. Presence of esophagitis > Los Angeles grade A classification
5. Presence of conditions precluding histological sampling of the esophagus (e.g., esophageal varices, coagulation disorders, anticoagulant therapy)
6. Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with barrett's esophagus or esophageal cancer referred for endoscopy
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-12; Primary Completion 2010-02 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
1. The number of patients and the number of lesions with HGD or early ACA detected with WLE and ETMI 2. The number of patients with HGD and early ACA detected with targeted biopsies only with ETMI and WLE | 2 years

SECONDARY OUTCOMES:
1. The positive predictive value (PPV) of HRE and AFI 2. The reduction of false-positive findings after NBI (both the initial in vivo NBI assessment as well as later assessment based on still images) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Louis M WongKeeSong, MD, Principal Investigator — Mayo Clinic
Locations (2):
- Mayo Clinic, Jacksonville, Florida, United States
- Academic Medical Center, Amsterdam, Netherlands